CLINICAL TRIAL: NCT01252147
Title: Inter-rater and Intra-rater Reliability Study of the Global Eyelash Assessment Scale for Assessment of Overall Eyelash Prominence
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 192024-066
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Results first posted 2012-09-28 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No treatment — No treatment (intervention) will be provided in this study

SUMMARY:
This study will evaluate the inter-rater and intra-rater reliability of the Global Eyelash Assessment (GEA) scale with photonumeric guide in Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to remove all eye makeup and facial jewelry during study

Exclusion Criteria:

* Permanent eyelid makeup or eyelash implants of any kind
* Eyelash tint or dye application within 2 months
* Eyelash extensions within 3 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Japanese adults
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2010-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Ueno, Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 68
Completed | 68
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 68
Age Continuous [Median (Full Range); unit: years] | 34.0 [20 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Overall Inter-Rater Reliability of Assessing Overall Eyelash Prominence Using the Japanese Global Eyelash Assessment Scale (GEA-J) at Day 1
Description: Inter-rater agreement (among raters) of the GEA-J scores (1=minimum,2=moderate, 3=marked, 4=very marked) to assess eyelash prominence was evaluated using Kendall's coefficient of concordance (Kendall's W). Each of 7 raters who scored 68 subjects' eyelashes using GEA-J Scale with photonumeric guide at 2 different time points at day 1. The overall inter-rater agreement for Kendall's W for all raters combined was estimated based on the average of the scores from those 2 different time points. The degree of agreement of the point estimates of Kendall's W was interpreted according to the reference range scale that was pre-defined as: <=0: poor, 0.00-0.20: slightly, 0.21-0.40: fair, 0.41-0.60: moderate, 0.61-0.80: substantial, 0.81-1:00: almost perfect. The 95% confidence interval for Kendall's W is provided.
Time Frame: Day 1
Population: Enrolled population, defined as all patients who were enrolled in (started) the study.
Measure: Number (95% Confidence Interval); unit: Kendall's W
Arm/Group | All Participants
Number analyzed (Participants) | 68
Kendall's W | 0.891 [0.653 to 1.000]

2. Primary Outcome: Overall Intra-Rater Reliability of Assessing Overall Eyelash Prominence Using the Japanese Global Eyelash Assessment Scale (GEA-J) at Day 1
Description: Intra-rater (within raters) agreement of the GEA-J scores (1=minimum, 2=moderate, 3=marked, 4=very marked) to assess eyelash prominence was evaluated by weighted Kappa statistics. Weighted Kappa statistics were calculated for each of 7 rater who evaluated 68 subjects using GEA-J scale with photonumeric guide, assessing agreement between 2 different time points at day 1. The overall intra-rater agreement for Kappa statistics for all raters combined was estimated by pooling Kappa statistics for each rater using a chi-square statistic. The degree of agreement of the point estimates of Kappa statistics was interpreted according to the reference range scale that was pre-defined as: <=0: poor, 0.00-0.20: slightly, 0.21-0.40: fair, 0.41-0.60: moderate, 0.61-0.80: substantial, 0.81-1:00: almost perfect. The 95% confidence interval for Kappa statistics is provided.
Time Frame: Day 1
Population: Enrolled population, defined as all patients who were enrolled in (started) the study.
Measure: Number (95% Confidence Interval); unit: Kappa statistics
Arm/Group | All Participants
Number analyzed (Participants) | 68
Kappa statistics | 0.818 [0.785 to 0.850]

ADVERSE EVENTS:
Description: Adverse event data were not collected/assessed.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo